CLINICAL TRIAL: NCT03962946
Title: Distal Radius Fracture: Clinical Outcome After Conservative Treatment in the Elder Patient
Acronym: RaDiX
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-00360; ch19Rikli2
Record Dates: First submitted 2019-05-22; First posted 2019-05-24 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Distal Radius Fracture
Keywords: Adolfsson-score; Suhm Score
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires to assess Patient reported Outcomes — Adolfsson-Score questionnaire quantifies the patient's utility of the hand. Suhm Score questionnaire quantifies the independency of a patient in his daily life.
Other: wrist function test — wrist function assessed by the range of motion (ROM) for both the affected and the unaffected side.

SUMMARY:
This study is performed to evaluate the outcome of conservative treatment after distal radius fractures in patients of 65 years or older at the time of the injury, primarily with respect to the prognostic value of the Adolfsson-score for the functional demands of the patient on his hand.

ELIGIBILITY:
Inclusion Criteria:

* Distal radius fracture with conservative treatment
* Treated in 2014 or 2015
* X-ray of injury
* Informed consent by the patient to participate in the study

Exclusion Criteria:

* No X-ray
* No signed informed consent
* Demented patients

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with a distal radius fracture who had undergone a conservative treatment at the University Hospital in Basel
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
Adolfsson score | single time point assessment at baseline
  Adolfsson-Score quantifies the patient's utility of the Hand; 8-point scale ranging from 1 = no activity done using hand/arm to 8 = professional activity with high physical stress for the arm. Lower scores reflect fewer effort in using arm/Hand; higher scores reflect higher strain in using arm/hand

SECONDARY OUTCOMES:
Suhm Score | single time point assessment at baseline
  Suhm Score quantifies the independency of a patient in his daily life. 4-point scale ranging from 1 = living at home, independent to 4 = living in nursing home, dependency. Lower scores reflect high independency of a patient in his daily life; higher scores reflect higher dependency of a patient in his daily life.
Quick Disabilities of the Arm, Shoulder and Hand (DASH) score | single time point assessment at baseline
  Quick DASH score is a 11-item, self-report questionnaire that measures physical function and symptoms in people with musculoskeletal disorders of the upper limb. The QuickDASH is scored in two components: the disability/symptom section (11 items, scored 1-5) and the optional high performance sport/Music or work modules (4 items, scored 1-5). A higher score indicates greater disability.
Range of wrist joint motion (degree) | single time point assessment at baseline
  Range of wrist joint motion (degree)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rikli, PD Dr. med, Principal Investigator — Department of Orthopaedic Surgery and Traumatology, University Hospital Basel
Locations (1):
- Department of Orthopaedics and Traumatology, University Hospital Basel, Basel, Switzerland